CLINICAL TRIAL: NCT03134014
Title: Long-term Effects of Consuming a High Protein, Beef Breakfast on Weight Management and Glycemic Control in Overweight 'Breakfast-skipping' Young People
Brief Title: High Protein Breakfast on Weight Management and Glycemic Control in 'Breakfast-skipping' Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Heather Leidy, Associate Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1611018501
Record Dates: First submitted 2017-04-19; First posted 2017-04-28 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Breakfast; Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior | interventions — Breakfast

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breakfast Skipping (BS) (No Intervention): The BS group will continue to skip breakfast.
- Normal Protein Breakfast (NP) (Active Comparator): The NP groups will be provided with the respective breakfast meals to consume, at home, between 6:00-8:00 am each day over the 4-mo intervention. The energy content of the breakfast meals will be standardized to 350 kcal. The NP breakfasts will be 11% protein (10 g protein), 63% CHO, and 26% fat
  Interventions: Dietary Supplement: Breakfast
- High Protein Breakfast (HP) (Active Comparator): The HP group will be provided with the respective breakfast meals to consume, at home, between 6:00-8:00 am each day over the 4-mo intervention. The energy content of the breakfast meals will be standardized to 350 kcal. The HP breakfasts will be 34% protein (30 g protein), 40% CHO, and 26% fat.
  Interventions: Dietary Supplement: Breakfast

INTERVENTIONS:
Dietary Supplement: Breakfast — If randomized to a breakfast consuming group, participants will be given breakfasts to consume between 6:00-8:00 am.
  Arms: High Protein Breakfast (HP); Normal Protein Breakfast (NP)

SUMMARY:
75 overweight, habitual 'breakfast-skipping' adolescents will complete the following long-term, randomized controlled trial. Participants will be randomly assigned to the following breakfast treatments: 350 kcal high protein breakfasts containing 30 g protein (primarily from lean beef), 35 g carbohydrates, and 10 g fat; 350 kcal normal protein breakfasts containing 10 g protein, 55 g carbohydrates, and 10 g fat; or will continue to skip breakfast. The following outcomes will be assessed during baseline and 4-month (post-intervention): body weight & body composition; waist circumference; daily food intake; 24-h free-living glycemic control; and pre and post-prandial satiety. In addition, body weight and free-living breakfast intake (quantity, quality, and type) will also be assessed at 2-month follow-up

DETAILED DESCRIPTION:
The NP and HP groups will be provided with their respective breakfast meals to consume, at home, between 6:00-8:00 am each day over the 4-mo intervention. The energy content of the NP and HP breakfast meals will be standardized to 350 kcal. The energy content of the breakfast meals is ~18% of daily energy intake estimated from the energy expenditure equations specific for adolescents ages 13-16 y. The NP breakfasts will be 11% protein (10 g protein), 63% CHO, and 26% fat, whereas the HP breakfasts will be 34% protein (30 g protein), 40% CHO, and 26% fat. The types of protein incorporated within the NP and HP meals will include a combination of beef (40%), dairy (20%), eggs (20%), and plant-based (20%) proteins. The NP and HP meals will include the same types of breakfasts but will vary in protein and CHO content. An 8-d breakfast rotation will occur throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. All ethnicities
3. Age: 15-21y
4. BMI/BMI Percentile: 20-34.0 kg/m2
5. Never smoked or used other tobacco products
6. Willing to consume the study breakfasts
7. Generally healthy (as assessed by Medical History Questionnaire)

Exclusion Criteria:

1. Clinically diagnosed with an eating disorder
2. Metabolic, hormonal, and/or neural conditions/diseases that influence metabolism or appetite
3. Currently or previously on a weight loss or other special diet (in the past 6 months)
4. Gained/lost ≥4.5kg over the past 6 months
5. Taking medication that would directly influence appetite (weight-loss drugs or antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months)

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Body Weight Change | Baseline and 4 months
  Body weight will be determined with a standard scale.
Body Composition Change | Baseline and 4 months
  Whole body total, fat, and fat free mass will be determined with DXA (GE) within the Bone and Body Composition Core of the Clinical Research Center. The DXA uses a linear X-ray fan beam with switched-pulse dual-energy and a multi-element detector array. The whole body scan takes <1.8 sec with radiation exposure of 0.01mGy. Waist circumference will be measured using a tape measure by one of the trained study staff members.
Energy Intake Change | Baseline and 4 months
  To assess the participant's total energy content all subjects will complete 3 dietary recalls over a 7-day period. The 3 days of data will be averaged together. Trained staff will contact the participant on 3 separate days (over a 7-day period) and ask questions related to the quantity, type, brand, preparation, and timing of food consumed throughout the previous day. Average energy intake will be assessed using the multi-pass system and NDSR (Nutrition Data System for Research). Change in energy intake(assessed as total energy content in kcal) will be determined.
24-h Free-Living Glycemic Control Change | Baseline and 4 months
  Free-living, glucose measures will be performed for 6 consecutive days using the Continuous Glucose Monitoring (CGM; Medtronic; Minneapolis, MN) used in our pilot study (1). The participants will report to our facility during the afternoon (on Day 1) for CGM insertion. A small area on the participant's abdomen will be cleaned and the tiny glucose sensor will be inserted just under the skin and held in place with tegaderm tape. The CGM measures glucose every 10sec and records an average glucose value every 5min for up to 144h. Calibration is performed by 4 finger sticks/d with a glucose analyzer.
Sleep Health Change | Baseline and 4 months
  Sleep health will be measured during 7 consecutive days through accelerometry/actigraphy (Actiwatch, Respironics; Philips, Pittsburgh PA). This device will be worn on the wrist, and the participants will continuously wear it over a 7-day period for measures of sleep quality.
Daily Appetite Change | Baseline and 4 months
  Questionnaires assessing the appetitive sensations (i.e., hunger, fullness, desire to eat, prospective food consumption), food cravings (sweet, savory-fat, meat), breakfast palatability (i.e., appearance, aroma, flavor, texture, overall liking), and perceived energy (sleepiness, energy, alertness) will be completed every waking hour for 3 days over a 7-day period. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The questionnaires will be completed on an iPod Touch using an in-house designed application (ScaleKit).
Food Craving Inventory Change | Baseline and 4 months
  Participants will fill out a Food Craving Inventory (FCI) questionnaire at baseline and 4-month (post-intervention). The FCI is a reliable and valid self-report measure of general and specific food cravings including cravings for high fat foods, carbohydrates/starches, sweets, and fast food (2). The FCI defines a craving as an intense desire to consume a particular food (or food type) that is difficult to resist. Further, this questionnaire prompts the participant to report how often (never, rarely, sometimes, often, always/almost every hour) he/she experienced a craving for the food throughout the day today.

SECONDARY OUTCOMES:
Body Weight (2-months post-intervention termination) Change | 5 months and 6 months
  Body weight will be determined with a standard scale.
Breakfast Intake (2-months post-intervention termination) Change | Average of 3 days at 6 months
  To assess the participant's energy content at breakfast, all subjects will complete 3 dietary recalls over a 7-day period and an average will of the 3 recalls will occur. Trained staff will contact the participant on 3 separate days (over a 7-day period) and ask questions related to the quantity, type, brand, preparation, and timing of food consumed throughout the previous breakfast meal. Breakfast energy content will be assessed using the multi-pass system and NDSR (Nutrition Data System for Research).

CONTACTS AND LOCATIONS:
Overall Officials: Heather Leidy, PhD, Principal Investigator — Associate Professor; Clinical Research Center (CTSI) Director
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauer LB, Reynolds LJ, Douglas SM, Kearney ML, Hoertel HA, Shafer RS, Thyfault JP, Leidy HJ. A pilot study examining the effects of consuming a high-protein vs normal-protein breakfast on free-living glycemic control in overweight/obese 'breakfast skipping' adolescents. Int J Obes (Lond). 2015 Sep;39(9):1421-4. doi: 10.1038/ijo.2015.101. Epub 2015 Jun 1. PMID 26028058
- [Background] White MA, Whisenhunt BL, Williamson DA, Greenway FL, Netemeyer RG. Development and validation of the food-craving inventory. Obes Res. 2002 Feb;10(2):107-14. doi: 10.1038/oby.2002.17. PMID 11836456